CLINICAL TRIAL: NCT05873608
Title: Communication Issues in Patient/Provider Discussions of Immunotherapy
Brief Title: Communication Issues in Patient and Provider Discussions of Immunotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rebecca D. Pentz, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00091198; NCI-2020-00828 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00091198; WINSHIP3293-16 (Other: Emory University Hospital/Winship Cancer Institute); P01CA257906 (NIH); P30CA138292 (NIH)
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Interviews as Topic; Observation; Watchful Waiting

STUDY DESIGN:
Intervention Model Description: For aim 4, each participant is assigned to watch a video and comprehension is tested using a pre and post method

ARMS (2):
- Interview (Other): Patients and providers undergo observation during a conversation about immunotherapy. Then participate in an interview over 20 minutes.
  Interventions: Other: Interview; Other: Observation
- Aim 4 tests an educational video (Other): The participants watch a video and their comprehension is tested in a pre and post methodology
  Interventions: Other: Educational video

INTERVENTIONS:
Other: Educational video — Testing an educational video
  Arms: Aim 4 tests an educational video
Other: Interview — Participate in interview
  Arms: Interview
Other: Observation — Undergo observation
  Other Names: Inspection; Visual Inspection
  Arms: Interview

SUMMARY:
This trials studies communication issues in patient and provider discussions about immunotherapy. The goal of this study is to describe where patients have heard about immunotherapy, what the participants understand about it, how physicians and other healthcare workers describe immunotherapy, and how educational videos may support patient knowledge about immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify misestimations about the risks and benefits of immunotherapy resulting from media hype or other sources and assess if these misestimations persist post-provider conversation about immunotherapy.

II. To qualitatively describe patient reported misunderstandings and to assess patient understanding of technical terms and metaphors used in the immunotherapy conversation.

III. To identify provider and patient preferences for information to be communicated about immunotherapy.

IV. Develop videos that describe immunotherapy and test their efficacy in improving understanding using pre and post methodology.

OUTLINE:

Patients and their providers undergo observation during a conversation about immunotherapy. Then participate in an interview over 20 minutes. Understanding of educational videos is then tested.

ELIGIBILITY:
Inclusion Criteria:

* AIMS 1-3: All patients and providers who may have a discussion about immunotherapy at the Winship Cancer Institute
* AIM 4: Any cancer patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2016-10-06 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2026-11-17 (Estimated)

PRIMARY OUTCOMES:
Misestimations about the risks and benefits of immunotherapy resulting from media hype or other sources | Up to 4 years
  Will use descriptive statistics to summarize the demographic characteristics and responses to the interviews. Will audio-record and transcribe the provider conversation for immunotherapy and the pre- and post-provider conversation interviews. The transcripts will be qualitatively coded using multi-level semantic analysis in MAXQDA. Pre-determined codes will include a list of potential benefits of immunotherapy, any patient estimation of the potential for benefit, any side effect and risk mentioned and any estimation of its frequency. Because there is no data on the frequency of misestimations due to media hype, no quantitative analysis is planned.
Qualitatively describe patient reported misunderstandings | Up to 4 years
  During the observed conversation, the ethics team member will note any technical term or metaphor used. The patient will then be asked if each term and metaphor is understood. The open ended questions about misunderstanding, technical terms and metaphors used, and patients' understanding of each term will be qualitatively coded using multi-level semantic analysis in MAXQDA. Frequency of misunderstood terms and misunderstood metaphors will be calculated.
Provider and patient preferences for information to be communicated about immunotherapy | Up to 4 years
  The frequencies of each item of information identified by providers and patients will be determined. A combined list of the most frequently mentioned items of information to be included and a discussion of immunotherapy will be compiled.
Correct definition rates (pre- versus post-video) | Up to 4 years
  Before-video and after-video correct definition rates will be calculated, along with 95% exact binomial confidence intervals using the Clopper-Pearson method. Before and after paired rates will be compared using an exact McNemar's test. Subset analyses will be performed for gender, age group (=< 55, > 55), and education level (high school graduate or less, some college or more).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Pentz, PhD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia